CLINICAL TRIAL: NCT05581225
Title: Prediction of Progression of Retinal Ischemia in Diabetes
Acronym: PREDICTION
Status: Active, not recruiting | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: 4C-029-22
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetes Mellitus (DM) is a major public health problem with significant socioeconomic implications due to its increased prevalence. Diabetic retinopathy (DR) is the most frequent complication in DM patients and remains the leading cause of legal blindness in working-age populations (Yau et al., 2012). Differentiating patients with higher vs low risk of progression to vision-threatening complications is of paramount importance for an efficient managing of the disease to prevent vision disability.

PREDICTION is a longitudinal prospective clinical study in DMT2 patients with a higher risk of progression to explore possible imaging, functional and systemic biomarkers of progression, using non-invasive methods, commonly applied in the clinical practice. Investigating the retinal vascular network (vessel density metrics with Optical Coherence Tomography Angiography) will allow a better understanding of the evolution of capillary closure and ischemia, two main risk factors for DR worsening.

DETAILED DESCRIPTION:
Patients with Mild to Severe NPDR (ETDRS DRSS 43-53) often progress to PDR and/or CI-DME (ETDRS Report). However, it is unclear which patients in this group are likely to progress. Previous studies have shown that diabetic macular ischemia (DMI) is a risk factor for progression of DR. This study aims to correlate baseline OCTA metrics with visual function and identify risk factors for progression from NPDR to PDR and/or CI-DME.

ELIGIBILITY:
Inclusion Criteria:

* DM type 2 according to 1985 WHO criteria.
* Age between 35 and 80 years.
* BCVA ≥ 75 letters (20 /32).
* Refraction with a spherical equivalent less than 5 Diopters.
* NPDR levels 43, 47 or 53 (based on the ETDRS criteria - 7 fields CFP).

Exclusion Criteria:

* Cataract or other eye disease that may interfere with fundus examinations.
* HBA1C ≥ 12%
* Any eye surgery within a period of 6-months before the inclusion visit date.
* Other retinal vascular disease.
* Previous laser or intravitreal injection treatment.
* Dilatation of the pupil < 5 mm.

Ages: 35 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 52 eyes from 52 individuals with T2D and NPDR with ETDRS DRSS grade 43, 47 or 53, with or without previous treatment, will be included in this study, in a recruitment period of 14 months.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
One and 2-steps change on ETDRS severity level (using standard 7-fields CFP acquisitions at 30º and in Wide-field 100º acquisitions). | 48 months
  Identify and characterize the progression of retinal microvascular changes (vascular occlusion) occurring in eyes with moderate to severe NPDR (ETDRS severity levels 43, 47 or 53).
Changes in Vessel density (VD) metrics (skeletonized VD, binarized VD (PD), considering macular region and midperiphery. | 48 months
  Explore new OCTA vascular metrics and identify which can be used as imaging biomarkers to better identify DR progression (skeletonized VD, binarized VD (PD).
Changes in geometric perfusion deficits (GPD) on the superficial and deep retinal vascular layers on SS-OCTA, considering macular region and midperiphery. | 48 months
  Explore new OCTA vascular metrics and identify which can be used as imaging biomarkers to better identify DR progression geometric perfusion deficits (GPD) using 3mm x 3mm and wide-field 15mm x 15mm OCTA acquisitions.

SECONDARY OUTCOMES:
Changes in FAZ area on OCTA | 48 months
Changes in perimeter on OCTA. | 48 months
Changes in circularity on OCTA. | 48 months
Changes in GCL + IPL thickness evaluated by SD-OCT. | 48 months
Changes in CRT and layer by layer thickness evaluated by SD-OCT. | 48 months
Changes in BCVA (ETDRS letters chart). | 48 months
Changes in mean luminous sensitivity in dB, evaluated by Microperimetry. | 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- AIBILI-CEC (AIBILI- Clinical Trials Centre), Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No